CLINICAL TRIAL: NCT07344480
Title: Retrospective Natural History Study of RASopathy-associated Cardiomyopathy
Acronym: RAS-CM
Status: Recruiting | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: RAS-CM
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-10

CONDITIONS: Hypertrophic Cardiomyopathy (HCM); Heart Failure; RASopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective data collection — Retrospective data collection, observation group are patients with genetic diagnosis of congenital RASopathy with hypertrophic cardiomyopathy and heart failure

SUMMARY:
RASopathy-associated hypertrophic cardiomyopathy (RAS-CM) is a disease with high morbidity and high mortality if presenting during infancy. Targeted therapies have shown significant activity in preclinical models and case reports. Drugs that target the underlying cause of this disease are now developed in cancer patients. Conducting randomized trials is not possible in severely ill infants with RAS-CM. Existing historical controls from older eras are not sufficient as external controls to support drug development as they lack critical clinical and genetic information to allow comparison with the cohort planned for future clinical trials.

The purpose of this investigator-initiated retrospective natural history study is to collect clinical information and genetic information in patients with RAS-CM. The first goal is to establish a data set that meets regulatory requirements for the use as external control data in a future clinical trial, composing non-randomized, single-arm, open-label study cohorts. The second goal is to obtain natural history information that supports the selection of secondary exploratory endpoints chosen in a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Molecular genetic diagnosis of a RASopathy (i.e., a pathogenic or likely pathogenic variant in one of the RAS-MAPK pathway genes identified, irrespective of when performed) AND Imaging diagnosis of myocardial hypertrophy (echocardiography) showing a maximal end-diastolic wall thickness of greater than normal (z-score > 2) with or without outflow tract obstruction AND Admitted to hospital between 01/01/2015 and 06/30/2019 for congestive heart failure* or developing progressive congestive heart failure during any hospital stay within first 6 months of life**

*Ross score calculated from medical history and physical examination notes in the absence of any other reason prompting hospital admission (e.g., elective procedure, other organ dysfunction, etc.); **: defined by Ross score greater than 2

Exclusion Criteria:

Receiving mTOR inhibitor and/or MEK inhibitors Inability to identify or retrospectively calculate the patient´s Ross score within the first six months of life

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To define the one-year transplant-free survival rate of patients with infantile-onset RASopathy-associated hypertrophic cardiomyopathy, admitted to the hospital with congestive heart failure by 6 months of age. | Admitted to hospital between 01/01/2015 and 06/30/2019 for congestive heart failure* or developing progressive congestive heart failure during any hospital stay within first 6 months of life**

CONTACTS AND LOCATIONS:
Locations (1):
- TUM Klinikum Deutsches Herzzentrum München, München, Germany